CLINICAL TRIAL: NCT03312699
Title: Effects of Aging on Primary and Secondary Vaccine Responses in a 15-Year Longitudinal Cohort
Brief Title: Effects of Aging on Primary and Secondary Vaccine Responses
Acronym: SLVP033
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Philip Grant, Assistant Professor of Medicine (Infectious Diseases), Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 40216; R01AI130398-01 (NIH)
Record Dates: First submitted 2017-10-12; First posted 2017-10-18 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Influenza; Hepatitis A; Typhoid; Healthy Adults
Keywords: Inactivated, quadrivalent influenza vaccine; Inactivated Hepatitis A vaccine; Inactivated, trivalent high-dose influenza vaccine; Typhoid Vi Polysaccharide Vaccine; Typhoid Vaccine Live Oral Ty21a; Influenza Vaccine, Adjuvanted
MeSH Terms: conditions — Influenza, Human; Hepatitis A; Typhoid Fever | interventions — Fluzone High-Dose; fluad vaccine; Hepatitis A Vaccines; Vi polysaccharide vaccine, typhoid; Ty21a typhoid vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Group A IIV4 (Experimental): Group A: Up to 30 healthy volunteers 18-40 years old, will be given seasonal quadrivalent inactivated influenza vaccine (IIV4) Fluzone® Quadrivalent vaccine. Each volunteer will complete a total of 4 visits: Day 0 (pre-immunization), Day 6-8, Day 12-16, and Day 28+ 7 (post-immunization). All visits will consist of drawing blood for study assays and monitoring for serious adverse events (SAEs).
  Interventions: Biological: Fluzone® quadrivalent
- Group B High Dose IIV3 (Experimental): Group B: Up to 15 healthy volunteers 65 plus years old, will be given seasonal high dose trivalent inactivated influenza vaccine (Fluzone High Dose) Fluzone® high dose vaccine. Each volunteer will complete a total of 4 visits: Day 0 (pre-immunization), Day 6-8, Day 12-16, and Day 28+ 7 (post-immunization). All visits will consist of drawing blood for study assays and monitoring for serious adverse events (SAEs).
  Interventions: Biological: Fluzone High Dose
- Group B Fluad (Experimental): Group B: Up to 15 healthy volunteers 65 plus years old, will be given seasonal adjuvanted trivalent inactivated influenza vaccine Fluad®. Each volunteer will complete a total of 4 visits: Day 0 (pre-immunization), Day 6-8, Day 12-16, and Day 28+ 7 (post-immunization). All visits will consist of drawing blood for study assays and monitoring for serious adverse events (SAEs).
  Interventions: Biological: Fluad
- Group A Hepatitis A (HepA) (Experimental): Group A: Up to 30 healthy volunteers 18-40 years old, will be given inactivated Hepatitis A vaccine Vaqta® in year 1 of the study and a booster 12 months post primary Vaqta vaccination. Each volunteer will complete a total of 4 visits per vaccination: Day 0 (pre-immunization), Day 6-8, Day 12-16, and Day 28+ 7 (post-immunization). All visits will consist of drawing blood for study assays and monitoring for serious adverse events (SAEs).
  Interventions: Biological: Vaqta
- Group B Hepatitis A (Experimental): Group B: Up to 30 healthy volunteers 65 plus years old, will be given inactivated Hepatitis A vaccine Vaqta® in year 1 of the study and a booster 12 months post primary Vaqta vaccination. Each volunteer will complete a total of 4 visits per vaccination: Day 0 (pre-immunization), Day 6-8, Day 12-16, and Day 28+ 7 (post-immunization). All visits will consist of drawing blood for study assays and monitoring for serious adverse events (SAEs).
  Interventions: Biological: Vaqta
- Group A Typhoid VI (Experimental): Group A: Up to 15 healthy volunteers 18-40 years old, will be randomized to either Typhoid Vi Polysaccharide Vaccine (Typhoid VI), Typhim Vi®, or Typhoid Vaccine Live Oral Ty21a, Vivotif®. This arm represents those randomized to Typhoid VI. Each volunteer will complete a total of 4 visits: Day 0 (pre-immunization), Day 6-8, Day 12-16, and Day 28+ 7 (post-immunization). All visits will consist of drawing blood for study assays and monitoring for serious adverse events (SAEs).
  Interventions: Biological: Typhim Vi
- Group A Oral Typhoid (Experimental): Group A: Up to 15 healthy volunteers 18-40 years old, will be randomized to either Typhoid Vi Polysaccharide Vaccine, Typhim Vi®, or Typhoid Vaccine Live Oral Ty21a, Vivotif® (Oral Typhoid). This arm represents those randomized to Oral Typhoid. Each volunteer will complete a total of 4 visits: Day 0 (pre-immunization), Day 6-8 (from date of last oral dose), Day 12-16, and Day 28+ 7 (post-immunization). All visits will consist of drawing blood for study assays and monitoring for serious adverse events (SAEs).
  Interventions: Biological: Vivotif
- Group B Typhoid VI (Experimental): Group B: Up to 30 healthy volunteers 65 plud years old, will be given Typhoid Vi Polysaccharide Vaccine (Typhoid VI), Typhim Vi® vaccine. Each volunteer will complete a total of 4 visits: Day 0 (pre-immunization), Day 6-8, Day 12-16, and Day 28+ 7 (post-immunization). All visits will consist of drawing blood for study assays and monitoring for serious adverse events (SAEs).
  Interventions: Biological: Typhim Vi

INTERVENTIONS:
Biological: Fluzone® quadrivalent — IIV4 vaccine will be administered as a 0.5 mL dose, with a sterile, disposable syringe and needle by intramuscular (IM) injection into the deltoid muscle.
  Other Names: IIV4 inactivated influenza vaccine
  Arms: Group A IIV4
Biological: Fluzone High Dose — High Dose IIV3 vaccine will be administered as a 0.5 mL dose, with a sterile, disposable syringe and needle by IM injection into the deltoid muscle.
  Other Names: High Dose Trivalent, inactivated influenza vaccine (TIV)
  Arms: Group B High Dose IIV3
Biological: Fluad — Fluad vaccine will be administered as a 0.5 mL dose, with a sterile, disposable syringe and needle by IM injection into the deltoid muscle.
  Other Names: Adjuvanted Trivalent, inactivated influenza vaccine
  Arms: Group B Fluad
Biological: Vaqta — Vaqta vaccine will be administered as a 1 mL dose, with a sterile, disposable syringe and needle by IM injection into the deltoid muscle.
  Other Names: Inactivated Hepatitis A Vaccine
  Arms: Group A Hepatitis A (HepA); Group B Hepatitis A
Biological: Typhim Vi — Typhim Vi vaccine will be administered as a 0.5 mL dose, with a sterile, disposable syringe and needle by IM injection into the deltoid muscle.
  Other Names: Typhoid Vi Polysaccharide Vaccine
  Arms: Group A Typhoid VI; Group B Typhoid VI
Biological: Vivotif — One capsule is to be swallowed approximately 1 hour before a meal with a cold or luke-warm [temperature not to exceed body temperature, e.g., 37 °C (98.6 °F)] drink on alternate days, e.g., days 1, 3, 5 and 7.
  Other Names: Typhoid Vaccine Live Oral Ty21a
  Arms: Group A Oral Typhoid

SUMMARY:
The purpose of this study is to use an existing, unique clinical cohort: the longitudinal cohort of younger (21-40 years) and elderly (>65 years) subjects whose yearly influenza vaccine responses have been studied extensively since 2007, to gain molecular and cellular mechanistic insights into the impaired vaccine responses in the elderly.

DETAILED DESCRIPTION:
This is a phase I mechanistic study of sixty 21-40 and >65 year old adult volunteers who previously participated in vaccine studies with our program. All participation is by invitation only.

The volunteers will be enrolled into two groups. Group A: Up to 30 healthy adult volunteers age 21-40 who will be given seasonal quadrivalent inactivated influenza vaccine (IIV4) prior to flu season for each of 5 years. They will also be given an inactivated Hepatitis A vaccine in the spring of years 1 and 2. Each volunteer will complete a total of 4 visits for each immunization: Day 0 (pre-immunization), Day 6-8, Day 12-15, and Day 26-30 (post-immunization). All visits will consist of drawing blood for study assays and monitoring for serious adverse events (SAEs).

A subset of this group will be randomized to receive either a Typhoid Vi Polysaccharide Vaccine or Typhoid Vaccine Live Oral Ty21a vaccine in year 3. Each volunteer will complete a total of 4 visits for this immunization: Day 0 (pre-immunization), Day 6-8 post completion of injection or final oral dose, Day 12-15 and Day 26-30 (post-immunization). All visits will consist of drawing blood for study assays and monitoring for serious adverse events (SAEs).

Group B: Up to 30 healthy adult volunteers age 65 plus who will be randomized and given seasonal trivalent high dose inactivated influenza vaccine (IIV3) or trivalent adjuvanted trivalent inactivated influenza vaccine (Fluad) prior to flu season for each of 5 years. They will also be given an inactivated Hepatitis A vaccine in the spring of years 1 and 2 and aTyphoid Vi Polysaccharide Vaccine in year 3. Each volunteer will complete a total of 4 visits for each immunization: Day 0 (pre-immunization), Day 6-8, Day 12-15, and Day 26-30 (post-immunization). All visits will consist of drawing blood for study assays and monitoring for serious adverse events (SAEs).

A subset of subjects (with a target of 10 younger and 10 older subjects depending on health), will undergo bone marrow aspirates one or two years after typhoid vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Prior participant in either the Ellison cohort or another Stanford vaccine study with archived samples.
4. Male or female, aged 18-40 years or 65 years and older.
5. In good general health as evidenced by medical history.

Exclusion Criteria:

1. Prior off-study vaccination with the current season influenza vaccine for influenza vaccinations.
2. Allergy to egg or egg products
3. Allergy to vaccine components, including thimerosal
4. Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
5. Receipt of blood or blood products within the past 6 months of any study vaccination or planned receipt of blood products prior to completion of Day 28 post-immunization visit.
6. Receipt of inactivated vaccine 14 days prior to study vaccination or planned vaccination prior to Day 28 after study vaccination.
7. Receipt of live, attenuated vaccine within 60 days of study vaccination or planned vaccination prior to Day 28 after study vaccination.
8. Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment or planned blood donation prior to Day 28 after study vaccination.
9. Use of investigational agents within 30 days prior to enrollment or planned use of investigational agents prior to completion of all study visits.
10. Need for allergy immunizations (that cannot be postponed) between Days 0 and 28 post-immunization.
11. Pregnant or lactating woman for all but influenza vaccine. A woman who is pregnant or breastfeeding may be evaluated by the Protocol Director to determine if influenza vaccination would affect volunteer safety and may be included at the discretion of the investigator. Blood sample collection will be adjusted as necessary for volunteer safety (e.g. blood collection volume for a pregnant woman would follow the minimal risk guidelines of 50 ml in an 8 week period and collection may not occur more frequently than 2 times per week).
12. Any condition, which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
hemagglutination inhibition assay (HAI) titers | Day 0 to Day 28
  HAI titers measured at Days 0 and 28 for influenza.

SECONDARY OUTCOMES:
related AEs occurring during the 28 days post vaccination | Day 0 to Day 28 post-each immunization
  related AEs occurring during the 28 days post vaccination for each of the vaccination types (Influenza, Hepatitis A, Typhoid)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Boyd, MD, PhD, Principal Investigator — Stanford School of Medicine, Dept. of Pathology; Cornelia Dekker, MD, Principal Investigator — Stanford School of Medicine, Dept. of Pediatrics
Locations (1):
- Stanford LPCH Vaccine Program, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The NIH Human Immunology Project Consortium (HIPC) data repositories (ImmPORT) may store the results of the research assays results. Genetic data that is developed in this study may be made available to other researchers through the National Center for Biotechnology Information (NCBI) databases. Results from research assays will be labeled with a unique identification code and the volunteer identity (except for age) will not be disclosed.
Time Frame: De-identified data will be loaded into ImmPort following completion of all data analysis
Access Criteria: De-identified data will be publicly available through ImmPort

DOCUMENTS (1):
  • Informed Consent Form (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/99/NCT03312699/ICF_000.pdf